CLINICAL TRIAL: NCT03842553
Title: Rescuers at Risk: Posttraumatic Stress Symptoms Differ Among Police Officers, Fire Fighters, Ambulance Personnel, and Emergency and Psychiatric Nurses
Brief Title: Posttraumatic Stress Symptoms Among Rescuers at Risk
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: PTSD2014
Record Dates: First submitted 2019-02-04; First posted 2019-02-15 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Trauma; PTSD; Self Efficacy; Coping Skills; Suicidal Ideation
Keywords: PTSD; Trauma; Coping; Self Efficacy
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic; Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Police officers: Police officers from the cantonal police forces in Bern, Switzerland
  Interventions: Other: No Intervention: anonymous online survey
- Firefighters: Firefighters from the professional fire service of the Canton Bern, Switzerland
  Interventions: Other: No Intervention: anonymous online survey
- Ambulance personnel: Ambulance personnel of the Canton Bern, Switzerland
  Interventions: Other: No Intervention: anonymous online survey
- Emergency nurses: Emergency nurses of the Emergency Unit of the University Hospital of Bern, Switzerland
  Interventions: Other: No Intervention: anonymous online survey
- Psychiatric nurses: Psychiatric nurses of the University Hospital of Psychiatry, University of Bern, Switzerland
  Interventions: Other: No Intervention: anonymous online survey

INTERVENTIONS:
Other: No Intervention: anonymous online survey

SUMMARY:
This cross-sectional, anonymous online survey aims to examine how salient variables influence PTSS, well-being, and suicidal ideation across the following professions of rescue workers: firefighters, ambulance personnel, police officers, and emergency and psychiatric nurses. PTSS, coping strategies, well-being, suicidal ideation, previously experienced and work-related trauma, and self-efficacy were measured and analyzed using multiple regression and structural equation modeling.

DETAILED DESCRIPTION:
Employees of rescue and emergency services are at a risk of posttraumatic stress symptoms (PTSS) due to exposure to trauma and work-related stressors. Salient predictors for the development of PTSS among rescue workers have been identified; however, little is known about how predictors (e.g. coping strategies) differ among professions requiring repeated engagement in emergencies. The present survey examines how these variables influence PTSS, well-being, and suicidal ideation across different professions of rescue Workers using multiple regression and structural equation modeling.

ELIGIBILITY:
Inclusion Criteria:

Employee at the rescue or emergency services. The participation in the anonymous online study is voluntary and promoted by the department heads at the places of work corresponding to the studied professions. No ethical approval is needed as the survey was voluntary and anonymous and participants gave consent to use the data with their participation.

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees of rescue and emergency services in the canton Bern, Switzerland: - Firefighters of the canton Bern
  * Ambulance personnel of the canton Bern
  * Police officers of the canton Bern
  * Emergency nurses of the University Hospital of Bern
  * Psychiatric nurses of University Hospital of Psychiatry, Bern
Sampling Method: Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
PTSS-10 | at baseline
  Posttraumatic Stress Symptoms assessed with the Post Traumatic Symptom Scale, a self-rating scale used in screening and follow-up studies on catastrophe that measures the most common posttraumatic symptoms (sleep disorders, nightmares, fear of reminders, etc.)

SECONDARY OUTCOMES:
Well-being | at baseline
  Mental well-being assessed with the German version of the shortest General Health Questionnaire 12 (GHQ-12). Psychological distress and psychiatric disorders were assessed with the German Version of the Brief Symptom Inventory (BSI).
Suicidal Ideation | within the last 12 months before the survey
  Participants were asked if they had suicidal ideation in the 12 months prior to the questionnaire
Psychological distress and psychiatric disorders | at baseline
  German Version of the Brief Symptom Inventory (BSI). The 53-item self-report questionnaire measures symptoms of general psychopathology.

OTHER OUTCOMES:
Self-efficacy | at baseline
  Self-efficacy was measured using the General Perceived Self-Efficacy Scale, a 10-item self-report instrument for personality diagnostics based on Banduras's concept of perceived self-efficacy that measures the general optimistic competence expectation
Coping Strategies | at baseline
  5-point Likert scale, ranging from a score of 1, indicating "not helpful"; to 5, "very helpful." According to the operationalization of Coolidge, coping strategies were divided into three main subscales: I) problem-focused coping strategies, which was comprised of the subscales of "instrumental support" (getting help and advice from psychologic professionals) and "active job coping" (debriefing with operation team, supervisor, and work colleagues); II) dysfunctional coping strategies, which included "substance use" (alcohol or medication), "avoidance" (avoidance of situations and emotions associated with the stressful/traumatic situation), and "self-distraction" (turning to work or other activities to take the mind off the stressful situation); III) emotion-focused coping strategy (humor, getting emotional support from close friends, thinking about the positive aspects of the job).
The burden of stressful job-related circumstances | at baseline
  The burden of stressful job-related circumstances, such as dealing with situations including people (aggressive and violent people, dealing with deaths or suicide, threats, dealing with relatives, involvement of children) and job-related conditions (incorrect or wrong information about the emergency situation, shift work, time pressure). Participants stated if they had ever experienced a presented situation, and if so, whether the situation caused a light or heavy stress burden.
work-unrelated trauma | at baseline
  Number of previous experienced work-unrelated trauma
work-related trauma | at baseline
  Number of experienced trauma at work

CONTACTS AND LOCATIONS:
Overall Officials: Leila Soravia, Ph.D., Principal Investigator — University Hospital of Psychiatry, University of Bern
Locations (1):
- University Hospital of Psychiatry, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soravia LM, Schwab S, Walther S, Muller T. Rescuers at Risk: Posttraumatic Stress Symptoms Among Police Officers, Fire Fighters, Ambulance Personnel, and Emergency and Psychiatric Nurses. Front Psychiatry. 2021 Jan 19;11:602064. doi: 10.3389/fpsyt.2020.602064. eCollection 2020. PMID 33542696